CLINICAL TRIAL: NCT06837142
Title: A Drug-drug Interaction Study With TS-172 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS172-03-05
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Triazolam; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triazolam and TS-172 (part A) (Experimental)
  Interventions: Drug: Triazolam and TS-172
- TS-172 and itraconazole (part B) (Experimental)
  Interventions: Drug: TS-172 and itraconazole

INTERVENTIONS:
Drug: Triazolam and TS-172 — Oral single administration of triazolam 0.25 mg at single administration phase, followed by a oral single administration of triazolam 0.25 mg and TS-172 20 mg at concomitant administration phase
  Arms: Triazolam and TS-172 (part A)
Drug: TS-172 and itraconazole — Oral single administrtation of TS-172 20 mg at single administration phase, followed by a oral single administration of TS-172 and itoraconazole 200 mg at concomitant administration phase
  Arms: TS-172 and itraconazole (part B)

SUMMARY:
An open-label, single-center, single-sequence study to evaluate the drug-drud interaction between the CYP3A substrate triazolam and TS-172 (part A) and the potent CYP3A inhibitor itraconazole and TS-172 (part B) in healthy male subjects on their pharmacokinetics, safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy adult males whose age is >=18 and <40 years at the time of obtaining informed consent
* Subjects whose body mass index is >=18.5 and <25.0 at the screening test
* Subjects who are judged by a principal investigator or a sub-investigator to be eligible for participation in the study based on the results at the screening test and before administration of the drugs used in the study
* Subjects who have been informed of the clinical trial, understand the details of the trial, and give their written consent prior to participation in the trial

Exclusion Criteria:

* Subjects with medical history ineligible for participation in the study such as of respiratory, cardiovascular, gastrointestinal, hepatic, renal, urologic, endocrine, metabolic, hematologic, immunologic, dermatologic, neurologic, or psychiatric diseases
* Subjects with medical history of disease (e.g., stomach or intestinal ulcers) or surgery (e.g., gastrectomy, gastric bandage, gastric bypass) that may affect the absorption of the drugs used in the study
* Subjects who have been hospitalized with any treatment or undergone surgery within 12 weeks prior to receiving the drugs used in the study
* Subjects with medical history of drug allergies (limited to severe symptoms such as anaphylaxis) or significant allergic predispositions (e.g., asthma that requires treatment)
* Subjects who have used medications (including over-the-counter drugs) within 2 weeks prior to receiving the drugs used in the study

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum plasma concentration (Cmax) of unchanged form of triazolam | Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours after dosing
Part A: Area under the concentration-time curve (AUC) from time zero to time of the last quantifiable concentration of unchanged form of triazolam in plasma | Up to 24 hours postdose
Part A: Area under the concentration-time curve (AUC) from time zero extrapolated to infinite time of unchanged form of triazolam in plasma | Up to 24 hours postdose
Part B: Maximum plasma concentration (Cmax) of unchanged form of TS-172 and its metabolite | Pre-dose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours after dosing
Part B: Area under the concentration-time curve (AUC) from time zero to time of the last quantifiable concentration of unchanged form of TS-172 and its metabolite in plasma | Up to 48 hours postdose
Part B: Area under the concentration-time curve (AUC) from time zero extrapolated to infinite time of unchanged form of TS-172 and its metabolite in plasma | Up to 48 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No